CLINICAL TRIAL: NCT04927455
Title: Pilot Study to Evaluate Impact and Transferability of an Alcohol Focused Harm Reduction Support System Based on Mental Health Recovery Named IACA!
Brief Title: Pilot Study to Evaluate "Intégrer et Accompagner Les Consommations d'Alcool!" (IACA!)'s Impact and Transferability
Acronym: VITAE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/35
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Craving; Addiction, Alcohol; Alcoholism
Keywords: Public Health; Alcohol use and addiction; risk reduction; innovation; mental health recovering; Transferability; Viability; Pilot study
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Behavior, Addictive; Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In France, alcohol consumption is the second most common cause of so-called preventable cancers after tobacco. Since 2014, in the "Provence-Alpes-Côte d'Azur" (PACA) region, the association Santé! has been developing an innovative intervention to support people suffering from alcohol-related addiction. This intervention, called IACA! must therefore be evaluated on a larger scale before conclusions about its effectiveness can be drawn from a comparative trial.

This evaluation requires significant human and material resources. It is therefore recommended to first assess the transferability of IACA! in other care centers in a pilot study.

DETAILED DESCRIPTION:
In France, 11% of cancers in men and 4.5% of cancers in women are attributed to alcohol consumption. It is the second leading cause of so-called preventable cancers, accounting for 28,000 alcohol-related cancers out of 352,000 new cases of cancer affecting annually adults (over 30 years of age). Overall, alcohol is among the top 3 factors contributing to Disability-Adjusted life year (DALYs) in France in 2017. Some cancer risks can be quantified as early as one drink a day (oesophagus, oral cavity, pharynx and breast in women). However, the risks associated with alcohol consumption remain influenced by the quantities consumed. There is therefore an interest, particularly for consumers of the largest quantities, in reducing the quantities consumed. In Europe, while people who drink more than 60 g/d of alcohol for men and 40 g/d for women are estimated to represent only 16.1% of the population for men and 9.3% for women, they represent 87% and 82% of alcohol-related morbidity and mortality respectively. Subjects with addiction (or substance use disorders) have an increased risk of social harm (1.5 to 3 times that of alcohol users without addiction), a higher mortality (1.4 to 6.5 compared to the general population) with a life expectancy of 9 to 20 years shorter than that of the general population. Moreover, even if the quantities consumed are not a valid individual diagnostic criterion, studies show a strong association between the quantity consumed and the diagnosis of addiction. Finally, some studies suggest that the prevalence of secondary harm from alcohol use follows an exponential curve as a function of alcohol consumption.

Since 2014, in the PACA region, the association Santé! has been developing an intervention to support people suffering from alcohol-related addiction. This intervention, called IACA! (Integrating and supporting alcohol consumption), differs from the support provided during rehabilitation cures and aims to: fight against discrimination and exclusion of people who drink alcohol, re-engage these individuals in the care process (because they have generally left it) by using the appropriate levers, promote well-being, improve quality of life and recovery and support the recovery in control of consumption. Thus, IACA!, through its philosophy and implementation, is based both on the risk reduction approach historically deployed with drug users and on the recovery approach, developed in the field of mental health. The first one-year results of this program were promising since, of 17 people who received the intervention, all had a social or health benefit, 13 of whom were associated with stabilization (n=4), reduction (n=7) or cessation (n=2) of alcohol use.

These promising results must therefore be evaluated on a larger scale before conclusions about its effectiveness can be drawn from a comparative trial. This type of evaluation requires significant human and material resources. It is therefore recommended to first assess in the field: 1) the conditions under which such an intervention is deployed in other centres (adaptations implemented by other centres to deploy IACA! for example, without distorting the intervention), 2) the acceptability and feasibility of the intervention in other centres (are the human and material resources on site sufficient for the successful deployment of the intervention?), 3) the acceptability and feasibility of the large-scale evaluation envisaged.

ELIGIBILITY:
Inclusion criteria common to the 3 populations:

* Over 18 years of age
* whatever the gender
* Non-opposition to participate

Inclusion criteria for professionals from centers implementing IACA! :

Concerning professionals in contact with the patients:

* Having been trained at IACA!
* Working in the centers participating in the implementation of IACA!

Concerning the persons in charge of the centers :

These professionals are those who have participated in the deployment of the IACA! method in their centers

Criteria for the inclusion of health professionals ! Participating or having recently participated in the implementation of IACA!

Exclusion Criteria:

The beneficiaries will be excluded if they have a severe somatic or psychiatric pathology that is incompatible with understanding the assessment tools; difficulty understanding and/or writing French; if they are unreachable by telephone, if they are participating in another research project with an ongoing exclusion period, if they are placed under court protection and if they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research will investigate three types of populations:
  * Individuals receiving support from the IACA! Intervention (called beneficiaries),
  * Professionals implementing the IACA! Intervention i.e. the pairs in charge of accompanying the beneficiaries in the centers as well as the persons in charge of these centers,
  * Professionals from Santé! supporting the deployment of the IACA! intervention.
  The beneficiaries are all persons integrating the program in the project's partner sites and consuming alcohol.
  The professionals will be specialized educators, social workers, nurses, social and solidarity economy advisors, etc.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Severity of alcohol use | 12 months after the start of IACA

SECONDARY OUTCOMES:
Utility dimension of viability - alcohol consumption | Baseline (M0)
  Average number of units of alcohol consumption in the past 30 days
Utility dimension of viability - alcohol consumption | 3 months (M3)
  Average number of units of alcohol consumption in the past 30 days
Utility dimension of viability - alcohol consumption | 6 months (M6)
  Average number of units of alcohol consumption in the past 30 days
Utility dimension of viability - alcohol consumption | 9 months (M9)
  Average number of units of alcohol consumption in the past 30 days
Utility dimension of viability - alcohol consumption | 12 months (M12)
  Average number of units of alcohol consumption in the past 30 days
Utility dimension of viability - craving | Baseline (M0)
  Craving: average frequency and intensity in the last 30 days
Utility dimension of viability - craving | 3 months (M3)
  Craving: average frequency and intensity in the last 30 days
Utility dimension of viability - craving | 6 months (M6)
  Craving: average frequency and intensity in the last 30 days
Utility dimension of viability - craving | 9 months (M9)
  Craving: average frequency and intensity in the last 30 days
Utility dimension of viability - craving | 12 months (M12)
  Craving: average frequency and intensity in the last 30 days
Utility dimension of viability - severity | Baseline (M0)
  Severity score for addictive substances and behaviors
Utility dimension of viability - severity | 3 months (M3)
  Severity score for addictive substances and behaviors
Utility dimension of viability - severity | 6 months (M6)
  Severity score for addictive substances and behaviors
Utility dimension of viability - severity | 9 months (M9)
  Severity score for addictive substances and behaviors
Utility dimension of viability - severity | 12 months (M12)
  Severity score for addictive substances and behaviors
Utility dimension of viability - disorders | Baseline (M0)
  Presence of alcohol and other substance use disorders (past 12 months and past)
Utility dimension of viability - disorders | 3 months (M3)
  Presence of alcohol and other substance use disorders (past 12 months and past)
Utility dimension of viability - disorders | 6 months (M6)
  Presence of alcohol and other substance use disorders (past 12 months and past)
Utility dimension of viability - disorders | 9 months (M9)
  Presence of alcohol and other substance use disorders (past 12 months and past)
Utility dimension of viability - disorders | 12 months (M12)
  Presence of alcohol and other substance use disorders (past 12 months and past)
Utility dimension of viability - Other substances | Baseline (M0)
  Number of days of use of other substances/behaviours in the past 30 days
Utility dimension of viability - Other substances | 3 months (M3)
  Number of days of use of other substances/behaviours in the past 30 days
Utility dimension of viability - Other substances | 6 months (M6)
  Number of days of use of other substances/behaviours in the past 30 days
Utility dimension of viability - Other substances | 9 months (M9)
  Number of days of use of other substances/behaviours in the past 30 days
Utility dimension of viability - Other substances | 12 months (M12)
  Number of days of use of other substances/behaviours in the past 30 days
Utility dimension of viability - Inventory | Baseline (M0)
  Inventory of medical, psychosocial and psycho-educational contacts in the last 30 days
Utility dimension of viability - Inventory | 3 months (M3)
  Inventory of medical, psychosocial and psycho-educational contacts in the last 30 days
Utility dimension of viability - Inventory | 6 months (M6)
  Inventory of medical, psychosocial and psycho-educational contacts in the last 30 days
Utility dimension of viability - Inventory | 9 months (M9)
  Inventory of medical, psychosocial and psycho-educational contacts in the last 30 days
Utility dimension of viability - Inventory | 12 months (M12)
  Inventory of medical, psychosocial and psycho-educational contacts in the last 30 days
Utility dimension of viability - QoL | Baseline (M0)
  Quality of life
Utility dimension of viability - QoL | 3 months (M3)
  Quality of life
Utility dimension of viability - QoL | 6 months (M6)
  Quality of life
Utility dimension of viability - QoL | 9 months (M9)
  Quality of life
Utility dimension of viability - QoL | 12 months (M12)
  Quality of life
Conditions of transferability | 9 to 12 months (M9 to M12)
  Conditions of transferability linked to the characteristics of the stakeholders and the context: contextual conditions for success within the centres, the characteristics of professionals and patients influencing outcomes
Viability and implementation | 6 to 12 months (M6 to M12)
  Implementation of IACA! (process, resources, activities) including the respect of IACA! success principles (skills, postures)
Viability and utility | 6 to 12 months (M6 to M12)
  "utility" dimension (as a complement to the secondary criteria) of viability through the recovery mechanisms identified as successful mental health recovery
Viability and affordability | 6 to 12 months (M6 to M12)
  Affordability for professionals and beneficiaries (financial, geographical, social and cultural levers and brakes of the intervention)
Viability and evaluability | 6 to 12 months (M6 to M12)
  Evaluability of IACA: carrying out this evaluation, the availability of professionals and beneficiaries to answer questionnaires and interviews, missing data in the questionnaires etc.
Viability and adaptability | 6 to 12 months (M6 to M12)
  Adaptability of IACA! (integration of the action into the context and the current organisation of the centres)
Viability and acceptability | 6 to 12 months (M6 to M12)
  Acceptability of IACA! by professionals and beneficiaries
Feasibility study capacity | 12 months (M12)
  The centres' capacity for inclusion (eligibility, recruitment rate, refusal rate)
Feasibility study complicance | 12 months (M12)
  The compliance rates; understanding, acceptability and feasibility of study questionnaires and data collection tools;
Feasibility study ressources | 12 months (M12)
  The ressources required (time required to complete all study forms, professional/centre capacity, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Cambon, PhD, Study Chair — Bordeaux University Hospital, Bordeaux University U1219; François Alla, MD, PhD, Study Director — Bordeaux University Hospital, Bordeaux University U1219; Marc Auriacombe, MD, PhD, Study Director — CNRS USR 3413 SANPSY, Bordeaux University, Bordeaux Hospital University
Locations (2):
- France (2):
  - CH Perrens - Equipe Addiction, Bordeaux
  - MéRISP - Université U1219, Bordeaux

REFERENCES:
- [Background] Thabane L, Cambon L, Potvin L, Pommier J, Kivits J, Minary L, Nour K, Blaise P, Charlesworth J, Alla F; Discussion Panel. Population health intervention research: what is the place for pilot studies? Trials. 2019 May 30;20(1):309. doi: 10.1186/s13063-019-3422-4. PMID 31146768
- [Background] Cambon L, Minary L, Ridde V, Alla F. Transferability of interventions in health education: a review. BMC Public Health. 2012 Jul 2;12:497. doi: 10.1186/1471-2458-12-497. PMID 22747988
- [Derived] Martin-Fernandez J, Stevens N, Moriceau S, Serre F, Blanc H, Latourte E, Auriacombe M, Cambon L. Realist evaluation of the impact, viability and transferability of an alcohol harm reduction support programme based on mental health recovery: the Vitae study protocol. BMJ Open. 2022 Aug 11;12(8):e065361. doi: 10.1136/bmjopen-2022-065361. PMID 35953259